CLINICAL TRIAL: NCT01046773
Title: Vitamin D Supplementation as Non-toxic Immunomodulation in Children With Crohn's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of California, Los Angeles (Other)
Collaborators: The Broad Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IBD-0285
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Crohn's Disease; Vitamin D Deficiency
Keywords: Children; Crohn's disease; Vitamin D
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Children with Crohn's disease less than 35 kg (Active Comparator): These are children ages 8 to 18 years inclusive, with mild to moderately active Crohn's disease.
  Interventions: Drug: Cholecalciferol
- Children with Crohn's disease 35 kg or greater (Active Comparator): These are children ages 8 to 18 years inclusive, with mild to moderately active Crohn's disease.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Children less than 35 kg will receive 2,000 IU oral cholecalciferol daily for 6 months.
  Arms: Children with Crohn's disease less than 35 kg
Drug: Cholecalciferol — Children 35 kg or greater will receive 4,000 IU oral cholecalciferol daily for 6 months.
  Arms: Children with Crohn's disease 35 kg or greater

SUMMARY:
IBD is caused by an abnormal immune response to the gut bacteria in people who are genetically predisposed. There has been a huge increase in the number of people diagnosed with IBD since World War II, likely due to changes in our environment. It is possible that the abundance of vitamin D in the body may be one of those environmental factors that the investigators can control to make patients with IBD better.

Vitamin D acts on cells of the immune system and causes many effects, including the production of a "natural antibiotic" called cathelicidin. The investigators know that when people are supplemented with vitamin D, levels of cathelicidin produced by these immune cells increase. By supplementing children with Crohn's disease with vitamin D, the investigators may be able to alter their immune system "naturally," making their disease better. A consensus of vitamin D experts believes that vitamin D levels need to reach a level of 40-70 ng/mL in the blood in order to have effects on the immune system. Raising vitamin D levels to this range is one of the goals in the current study.

DETAILED DESCRIPTION:
Vitamin D is an important nutrient controlling the health and development of our bones. Many patients with inflammatory bowel disease (IBD) are deficient in levels of vitamin D in their bodies. This is probably because vitamin D is lost from inflamed intestinal tissue into the stools. But while much attention has been given to studying the impact of vitamin D deficiency on the bone status of patients with IBD, our understanding of how vitamin D deficiency might affect the immune system in these patients is relatively poor.

The investigators intend to study vitamin D supplementation in children with Crohn's disease, ages 8 to 18 years. At the time of enrollment, the investigators will gather data on disease activity using both a simple history and physical exam, as well as blood and stool tests. In addition, the investigators will measure the levels of cathelicidin produced by the immune cells in their blood. The investigators will then supplement 20 children with vitamin D for a total of 6 months. During the study, patients will be seen every two months, where the investigators will monitor their vitamin D levels as well as perform rigorous safety monitoring for toxicity using blood and urine tests.

And at study conclusion, the investigators will again judge their disease severity and check their vitamin D levels in addition to tests of cathelicidin levels. The investigators believe that at study conclusion, the investigators will have achieved several important objectives. First, as a public health benefit, the investigators will show that large doses of supplemental vitamin D are safe in children and provide more benefit with less risk. Our patients will achieve those levels of vitamin D agreed by expert opinion that are required to cause effects on the immune system, and the investigators will see an increase in the amount of cathelicidin produced by their immune cells. As an added piece of information, the investigators would like to determine if there are any improvements in disease activity in patients supplemented with vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate Crohn's disease
* 8 to 18 years old, inclusive

Exclusion Criteria:

* Children less than 8 years or greater than 18 years at the time of study screening
* Patients with a documented history of hypercalcemia, renal insufficiency, or nephrolithiasis
* Patients taking cholestyramine
* Patients who have a GI tract in discontinuity (ostomy)
* Patients who have serum 25-OH vitamin D levels of >50 ng/mL at the time of study screening

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The investigators aim to achieve patient target serum levels of 25-hydroxy vitamin D between 40-60 ng/mL after 6 months of supplementation | 6 months
The investigators aim to determine the association between vitamin D supplementation and cathelicidin production. | 6 months

SECONDARY OUTCOMES:
Detect changes in Crohn's disease activity: clinically, biochemically, and by surrogate markers. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ziring, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Pappa HM, Bern E, Kamin D, Grand RJ. Vitamin D status in gastrointestinal and liver disease. Curr Opin Gastroenterol. 2008 Mar;24(2):176-83. doi: 10.1097/MOG.0b013e3282f4d2f3. PMID 18301268
- [Background] Holick MF. The vitamin D deficiency pandemic and consequences for nonskeletal health: mechanisms of action. Mol Aspects Med. 2008 Dec;29(6):361-8. doi: 10.1016/j.mam.2008.08.008. Epub 2008 Sep 2. PMID 18801384
- [Background] Lo CW, Paris PW, Clemens TL, Nolan J, Holick MF. Vitamin D absorption in healthy subjects and in patients with intestinal malabsorption syndromes. Am J Clin Nutr. 1985 Oct;42(4):644-9. doi: 10.1093/ajcn/42.4.644. PMID 4050723
- [Background] Vogelsang H, Schofl R, Tillinger W, Ferenci P, Gangl A. 25-hydroxyvitamin D absorption in patients with Crohn's disease and with pancreatic insufficiency. Wien Klin Wochenschr. 1997 Sep 19;109(17):678-82. PMID 9331957
- [Background] Leichtmann GA, Bengoa JM, Bolt MJ, Sitrin MD. Intestinal absorption of cholecalciferol and 25-hydroxycholecalciferol in patients with both Crohn's disease and intestinal resection. Am J Clin Nutr. 1991 Sep;54(3):548-52. doi: 10.1093/ajcn/54.3.548. PMID 1652198
- [Background] Liu N, Nguyen L, Chun RF, Lagishetty V, Ren S, Wu S, Hollis B, DeLuca HF, Adams JS, Hewison M. Altered endocrine and autocrine metabolism of vitamin D in a mouse model of gastrointestinal inflammation. Endocrinology. 2008 Oct;149(10):4799-808. doi: 10.1210/en.2008-0060. Epub 2008 Jun 5. PMID 18535110
- [Background] Schauber J, Rieger D, Weiler F, Wehkamp J, Eck M, Fellermann K, Scheppach W, Gallo RL, Stange EF. Heterogeneous expression of human cathelicidin hCAP18/LL-37 in inflammatory bowel diseases. Eur J Gastroenterol Hepatol. 2006 Jun;18(6):615-21. doi: 10.1097/00042737-200606000-00007. PMID 16702850
- [Background] Tai EK, Wu WK, Wong HP, Lam EK, Yu L, Cho CH. A new role for cathelicidin in ulcerative colitis in mice. Exp Biol Med (Maywood). 2007 Jun;232(6):799-808. PMID 17526772
- [Background] Martineau AR, Wilkinson KA, Newton SM, Floto RA, Norman AW, Skolimowska K, Davidson RN, Sorensen OE, Kampmann B, Griffiths CJ, Wilkinson RJ. IFN-gamma- and TNF-independent vitamin D-inducible human suppression of mycobacteria: the role of cathelicidin LL-37. J Immunol. 2007 Jun 1;178(11):7190-8. doi: 10.4049/jimmunol.178.11.7190. PMID 17513768
- [Background] Froicu M, Weaver V, Wynn TA, McDowell MA, Welsh JE, Cantorna MT. A crucial role for the vitamin D receptor in experimental inflammatory bowel diseases. Mol Endocrinol. 2003 Dec;17(12):2386-92. doi: 10.1210/me.2003-0281. Epub 2003 Sep 18. PMID 14500760
- [Background] Simmons JD, Mullighan C, Welsh KI, Jewell DP. Vitamin D receptor gene polymorphism: association with Crohn's disease susceptibility. Gut. 2000 Aug;47(2):211-4. doi: 10.1136/gut.47.2.211. PMID 10896912
- [Background] Heaney RP. Lessons for nutritional science from vitamin D. Am J Clin Nutr. 1999 May;69(5):825-6. doi: 10.1093/ajcn/69.5.825. No abstract available. PMID 10232617
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Maalouf J, Nabulsi M, Vieth R, Kimball S, El-Rassi R, Mahfoud Z, El-Hajj Fuleihan G. Short- and long-term safety of weekly high-dose vitamin D3 supplementation in school children. J Clin Endocrinol Metab. 2008 Jul;93(7):2693-701. doi: 10.1210/jc.2007-2530. Epub 2008 Apr 29. PMID 18445674
- [Background] Adams JS, Ren S, Liu PT, Chun RF, Lagishetty V, Gombart AF, Borregaard N, Modlin RL, Hewison M. Vitamin d-directed rheostatic regulation of monocyte antibacterial responses. J Immunol. 2009 Apr 1;182(7):4289-95. doi: 10.4049/jimmunol.0803736. PMID 19299728
- [Background] Vieth R. Vitamin D toxicity, policy, and science. J Bone Miner Res. 2007 Dec;22 Suppl 2:V64-8. doi: 10.1359/jbmr.07s221. PMID 18290725